CLINICAL TRIAL: NCT02807376
Title: A Prospective, Randomized, Controlled, Multi-Center Evaluation of a Powered Vascular Stapler in Laparoscopic Nephrectomies and Nephroureterectomies
Brief Title: An Evaluation of a Powered Vascular Stapler in Laparoscopic Nephrectomies and Nephroureterectomies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ethicon Endo-Surgery (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-002
Record Dates: First submitted 2016-06-14; First posted 2016-06-21 (Estimated); Results first posted 2018-12-19 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-11

CONDITIONS: Excision of Kidney

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Surgeon's 'standard of care' stapler (Active Comparator): Surgeon's standard of care stapler
  Interventions: Device: Surgeon's 'standard of care' stapler
- Ethicon Powered Vascular Stapler (Experimental): Ethicon Powered Vascular Stapler
  Interventions: Device: Ethicon Powered Vascular Stapler

INTERVENTIONS:
Device: Surgeon's 'standard of care' stapler
  Arms: Surgeon's 'standard of care' stapler
Device: Ethicon Powered Vascular Stapler
  Arms: Ethicon Powered Vascular Stapler

SUMMARY:
This prospective, randomized, controlled, multi-center study will collect and compare data from the surgeon's current standard of care stapler (for renal artery and renal vein transection) and powered vascular stapler

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for a simple or radical laparoscopic nephrectomy or a laparoscopic nephroureterectomy in accordance with the institution's standard of care (SOC);
* Performance status 0-1 (Eastern Cooperative Oncology Group classification), if applicable;
* American Society of Anesthesiologists (ASA) score < 3;
* No prior history of partial or wedge nephrectomy (on the kidney in which the procedure will be performed);
* Willing to give consent and comply with study-related evaluation and treatment schedule; and
* At least 18 years of age

Exclusion Criteria:

* Prior chemotherapy or radiation (within 30 days prior to the procedure or the duration of the subject's enrollment);
* Pregnancy;
* Physical or psychological condition which would impair study participation; or
* The subject is judged unsuitable for study participation by the Investigator for any other reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2016-07-05 (Actual); Primary Completion 2017-08-23 (Actual); Study Completion 2017-08-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Emory University, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was from July 2016 to July 2017 across 11 hospitals.
Pre-assignment Details: In total, 302 subjects were screened, 270 subjects were randomized, and those 32 subjects who were not randomized did not satisfy inclusion or exclusion criteria.
Groups:
- Standard of Care: Facility's Current Instrumentation
- Powered Vascular Stapler: Use of the ECHELON FLEX™ Powered Vascular Stapler
Period: Overall Study
Arm/Group | Standard of Care | Powered Vascular Stapler
Started | 139 | 131
Completed | 136 | 130
Not Completed | 3 | 1
Not completed — Intra-operative exclusion criteria | 3 | 0
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care | Powered Vascular Stapler | Total
Number analyzed (Participants) | 139 | 131 | 270
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.1 (14.0) | 63.6 (13.8) | 63.8 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 60 | 128
  Male | 71 | 71 | 142
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 1 | 7
  Not Hispanic or Latino | 39 | 38 | 77
  Unknown or Not Reported | 94 | 92 | 186
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 13 | 11 | 24
  White | 119 | 116 | 235
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 2 | 7

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Vessels Transected Requiring Intra-Operative Hemostatic Interventions
Description: Proportion of hemostatic interventions/procedures completed for intra-operative bleeding related to the transection of the Reanl Artery and Renal Vein during laparoscopic nephrectomy or nephroureterectomy with the use of standard of care stapler (SOC) or powered vascular stapler (PVS) defined as bleeding detected and controlled intraoperatively (additional stapling, over-sewing, clip placement, compression, use of suture, sealant, and/or buttress, and/or use of energy); or bleeding that occurs intra-operatively requiring blood or blood product transfusion or an additional surgical procedure (e.g. conversion to open).
Time Frame: Intra-Operative, an average of 2.6 hours, ranging from 42 minutes to 6.4 hours
Population: All randomized subjects in whom the Standard of Care or Powered Vascular Stapler was used for vessel transection.
Measure: Number (95% Confidence Interval); unit: proportion of transected vessels
Units Other Than Participants: Vessels Transected
Arm/Group | Standard of Care | Powered Vascular Stapler
Number analyzed (Participants) | 139 | 131
Number analyzed (Vessels Transected) | 309 | 305
proportion of transected vessels | 0.1359 [0.0977 to 0.1741] | 0.1836 [0.1402 to 0.2271]

2. Secondary Outcome: Proportion of Participants Requiring Post-operative Interventions or Procedures Related to Renal Artery or Renal Vein Bleeding
Description: Proportion of participants with hemostatic interventions /procedures completed for post-operative bleeding related to the transection of the Renal Artery and Renal Vein during laparoscopic nephrectomy or nephroureterectomy with the use of SOC or PVS:
  * Hemostasis intervention: bleeding that occurs post-operatively requiring blood or blood product transfusion or an additional surgical procedure (related to Renal Artery and Renal Vein transection).
  No hemostasis intervention is defined as no interventions needed for post-operative bleeding (related to PA and PV transection).
Time Frame: Post-Op through 4 Week Follow-up
Population: All randomized subjects in whom the Standard of Care or Powered Vascular Stapler was used for vessel transection.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Standard of Care | Powered Vascular Stapler
Number analyzed (Participants) | 139 | 131
proportion of participants | 0.0144 [0.0 to 0.0342] | 0.0076 [0.0 to 0.0225]

ADVERSE EVENTS:
Time Frame: 4 Weeks Post Procedure
Arm/Group | Standard of Care | Powered Vascular Stapler
All-Cause Mortality (participants affected / at risk) | 0/139 | 0/131
Serious Adverse Events (participants affected / at risk) | 21/139 | 14/131
Other Adverse Events (participants affected / at risk) | 26/139 | 33/131
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard of Care (N=139) | Powered Vascular Stapler (N=131)
Anemia (Blood and lymphatic system disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 2 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 1 | 0
Retroperitoneal hematoma (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Chest pain (General disorders) | 1 | 0
Device occlusion (General disorders) | 0 | 1
Pain (General disorders) | 1 | 0
Abdominal sepsis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 2 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 2
Urosepsis (Infections and infestations) | 1 | 1
Wound infection (Infections and infestations) | 1 | 1
Post procedural hemmorrhage (Injury, poisoning and procedural complications) | 3 | 0
Post-operative ileus (Injury, poisoning and procedural complications) | 1 | 1
Procedural complication (Injury, poisoning and procedural complications) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Hematuria (Renal and urinary disorders) | 1 | 1
Genital pain (Reproductive system and breast disorders) | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Wound drainage (Surgical and medical procedures) | 0 | 1
Hematoma (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Standard of Care (N=139) | Powered Vascular Stapler (N=131)
Nausea (Gastrointestinal disorders) | 6 | 7
Vomiting (Gastrointestinal disorders) | 5 | 11
Pyrexia (General disorders) | 5 | 6
Urinary tract infection (Infections and infestations) | 4 | 6
Wound infection (Infections and infestations) | 6 | 6
Urinary retention (Renal and urinary disorders) | 3 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2015-11-17): https://cdn.clinicaltrials.gov/large-docs/76/NCT02807376/Prot_000.pdf
  • Statistical Analysis Plan (2017-10-11): https://cdn.clinicaltrials.gov/large-docs/76/NCT02807376/SAP_001.pdf